CLINICAL TRIAL: NCT07068763
Title: Node-Sparing Short-Course Radiation Combined With Capecitabine and PD-1/CTLA-4 for MSS Early Middle and Low Rectal Cancer (mRCAT-E): An Open-label, Single-arm, Prospective Multicenter Clinical Trial
Brief Title: Node-Sparing Short-Course Radiation Combined With Capecitabine and PD-1/CTLA-4 for MSS Early Rectal Cancer
Acronym: mRCAT-E
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sir Run Run Shaw Hospital (Other)
Responsible Party: Principal Investigator, Zhangfa Song, Vice president, Sir Run Run Shaw Hospital, Qingchun Campus, Zhejiang University School of Medicine,
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SRRS-mRCAT-E
Record Dates: First submitted 2025-07-07; First posted 2025-07-16 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Rectal Cancer
Keywords: lymph-node-sparing short-course radiotherapy; capecitabine; PD-1 inhibitor; CTLA-4 inhibitor; organ preservation; clinical complete response
MeSH Terms: conditions — Rectal Neoplasms | interventions — Capecitabine

STUDY DESIGN:
Intervention Model Description: Single-arm, open-label trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Experimental Arm (Experimental): Patients receive lymph-node-sparing short-course radiotherapy of 25 Gy delivered in five daily fractions to the primary tumor bed (no nodal fields). Beginning on treatment Day 8, patients receive capecitabine 1,000 mg/m² orally twice daily on Days 1-14 plus PD-1/CTLA-4 inhibitor (5 mg/kg IV every 3 weeks) for four cycles. Tumor response is assessed 1-2 weeks after the last cycle; patients with clinical complete response enter a watch-and-wait program, while non-responders proceed to local excision or total mesorectal excision.
  Interventions: Radiation: Lymph-node-sparing short-course radiotherapy; Drug: Capecitabine; Drug: PD-1/CTLA-4 inhibitor (Aiparolitoworixureli injection)

INTERVENTIONS:
Radiation: Lymph-node-sparing short-course radiotherapy — Three-dimensional conformal or intensity-modulated radiotherapy targeting only the primary tumor bed (no regional lymph nodes), delivering a total dose of 25 Gy in 5 Gy fractions over five consecutive days.
Drug: Capecitabine — Oral capecitabine 1,000 mg/m² administered twice daily on Days 1-14 of each 21-day cycle, for a total of four cycles.
Drug: PD-1/CTLA-4 inhibitor (Aiparolitoworixureli injection) — Intravenous PD-1/CTLA-4 bispecific monoclonal antibody at 5 mg/kg every 3 weeks for four cycles, starting on Day 8 after completion of radiotherapy.

SUMMARY:
This is a single-arm, prospective, multicenter study evaluating a novel neoadjuvant treatment strategy for patients with early, mid-low rectal adenocarcinoma that is microsatellite stable (MSS). Instead of irradiating regional lymph nodes, we deliver short-course radiotherapy (25 Gy in 5 fractions) exclusively to the primary tumor ("lymph-node-sparing" approach), immediately followed by four 3-week cycles of capecitabine plus combined PD-1/CTLA-4 immune checkpoint inhibitors. Two weeks after completing chemo-immunotherapy, tumor response is assessed. Patients who achieve a clinical complete response may enter a "watch-and-wait" program; others will undergo local excision or total mesorectal excision (TME) as appropriate. The primary endpoint is the rate of complete response (clinical and pathological). Secondary endpoints include organ-preservation rate, 3-year local recurrence, 3-year disease-free and overall survival, toxicity, and quality-of-life measures. Results from a pilot study suggest that this regimen may substantially improve complete response rates while reducing radiation-related toxicity, potentially allowing more patients to avoid radical surgery and permanent stoma.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have a strong willingness to preserve the anus and are willing to receive neoadjuvant therapy.
2. Male or Female aged 18-80.
3. Patients diagnosed with low rectal cancer within 7 cm from the lower edge of the tumor to the anal verge by pelvic MRI and rectal ultrasound, the clinical stage is cT2-3N0M0.
4. Histologically confirmed rectal adenocarcinoma; Genetic testing suggests MSI-L or MSS, or tumor biopsy immunohistochemistry reveals pMMR, that is, MSH1, MSH2, MSH6, and PMS2 are all positive.
5. Eastern Cooperative Oncology Group (ECOG) score 0-1.
6. No previous treatment (including anti-tumor therapy, immunotherapy or pelvic radiation).
7. Informed consent form signed.

Exclusion Criteria:

1. Patients with a previous history of malignant tumors besides rectal cancer.
2. Patients with distant metastases before enrollment.
3. Patients with metastatic regional or non-regional lymph nodes are assessed by MRI or CT.
4. Patients with obstruction, perforation, or bleeding that require emergency surgery.
5. Patients with severe concomitant diseases and estimated survival time ≤ 5 years.
6. Allergic to any component of the therapy.
7. Patients who received immunosuppressive or systemic hormone therapy for immunosuppressive purposes within 1 month prior to the initiation of therapy.
8. Contraindications to radiotherapy and chemotherapy.
9. Patients who have received any other experimental drug (including immunotherapy) or participated in another interventional clinical trial within 30 days before screening.
10. Factors leading to study termination, such as alcoholism, drug abuse, other serious illnesses (including psychiatric disorders) requiring combination therapy, and patients with severe laboratory abnormalities. Patients with congenital or acquired immune deficiency (such as HIV infection).
11. Vulnerable groups, including mentally ill, cognitively impaired, critically ill patients, minors, pregnant or lactating women, illiterate, etc.

    Other conditions that investigators consider not suitable for this study.
12. Patient not suitable for participating by other concerns of researchers.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2025-10-09 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical and pathological complete response rate (CR rate) | Up to 12 weeks after completion of chemo-immunotherapy
  Proportion of enrolled patients who achieve a clinical complete response (cCR) on imaging, endoscopy, and biopsy and/or a pathological complete response (pCR) in surgical specimens (if resected) following lymph-node-sparing short-course radiotherapy combined with capecitabine and PD-1/CTLA-4 inhibitor.

SECONDARY OUTCOMES:
Organ preservation rate | 1 year after enrollment
  Proportion of patients who avoid total mesorectal excision (TME) and permanent stoma by remaining in watch-and-wait or undergoing only local excision.
3-year local recurrence rate | 3 years
  Proportion with tumor recurrence in the pelvis
Overall survival(OS） | 3 years after chemotherapy or surgery
  The three-year overall survival of patients.
Adverse effects rate | From date of initiation of treatment until the date of death from any cause, assessed up to 3 years
  Rate of radiotherapy, chemotherapy and immunotherapy related adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Sir run run shaw hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Lezoche E, Guerrieri M, Paganini AM, D'Ambrosio G, Baldarelli M, Lezoche G, Feliciotti F, De Sanctis A. Transanal endoscopic versus total mesorectal laparoscopic resections of T2-N0 low rectal cancers after neoadjuvant treatment: a prospective randomized trial with a 3-years minimum follow-up period. Surg Endosc. 2005 Jun;19(6):751-6. doi: 10.1007/s00464-004-8930-x. Epub 2005 May 4. PMID 15868260
- [Result] Annals of Oncology (2024) 24 (suppl_1): 1-20. 10.1016/iotech/iotech100744
- [Result] Habr-Gama A, Perez RO, Wynn G, Marks J, Kessler H, Gama-Rodrigues J. Complete clinical response after neoadjuvant chemoradiation therapy for distal rectal cancer: characterization of clinical and endoscopic findings for standardization. Dis Colon Rectum. 2010 Dec;53(12):1692-8. doi: 10.1007/DCR.0b013e3181f42b89. PMID 21178866